CLINICAL TRIAL: NCT03569059
Title: Optimizing Hand Rehabilitation Post Stroke Using Interactive Virtual Environments
Brief Title: Robot Assisted Virtual Rehabilitation for the Hand Post Stroke (RAVR)
Acronym: RAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Jersey Institute of Technology (Other)
Collaborators: Rutgers University (Other); Northeastern University (Other); Kessler Foundation (Other)
Responsible Party: Principal Investigator, Sergei V. Adamovich PhD, Professor, New Jersey Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD058301 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-06-26 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Stroke, Acute
Keywords: Stroke; Virtual Environment; Robotics; Upper Extremity; Hand; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of four groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early Robotic/VR Therapy (EVR) (Experimental): Subjects in this group will receive state-of-art inpatient usual care therapy plus 10 days of extra 1-hour/day of intensive therapy focusing on the hand using haptic robots integrated with complex gaming and virtual environments and initiated 5-30 days post stroke.
  Interventions: Device: Early Robotic/VR Therapy (EVR)
- Delayed Robotic/VR Therapy (DVR) (Experimental): Subjects in this group will receive state-of-art usual care therapy (inpatient and outpatient) plus 10 days of extra 1-hour/day of intensive therapy focusing on the hand using haptic robots integrated with complex gaming and virtual environments and initiated within 31-60 days post stroke.
  Interventions: Device: Delayed Robotic/VR Therapy (DVR)
- Usual Physical Therapy Care (No Intervention): Subjects in this group will receive state-of-art usual physical therapy/occupational therapy care.
- Dose-Matched Usual Physical Therapy Care (Experimental): Subjects in this group will receive state-of-art usual physical therapy/occupational therapy care plus an extra hour of state-of-art usual care.
  Interventions: Behavioral: Dose-Matched Usual Physical Therapy Care

INTERVENTIONS:
Device: Early Robotic/VR Therapy (EVR) — Subjects will perform state-of-art inpatient usual care therapy. In addition, they will perform an extra 1-hour/day of intensive therapy focusing on the hand in the form of interactive virtual reality games while assisted by robots. This additional treatment will be initiated 5-30 days post stroke.
  Other Names: NJIT-RAVR, NJIT-TrackGlove
  Arms: Early Robotic/VR Therapy (EVR)
Behavioral: Dose-Matched Usual Physical Therapy Care — Subjects will perform state-of-art usual physical/occupational care and 10 days of one additional hour of state-of-art usual inpatient and/or outpatient physical therapy/occupational therapy.
  Arms: Dose-Matched Usual Physical Therapy Care
Device: Delayed Robotic/VR Therapy (DVR) — Subjects will perform state-of-art inpatient usual care therapy. In addition, they will perform an extra 1-hour/day of intensive therapy focusing on the hand in the form of interactive virtual reality games while assisted by robots. This additional treatment will be initiated 31-60 days post stroke.
  Other Names: NJIT-RAVR, NJIT-TrackGlove
  Arms: Delayed Robotic/VR Therapy (DVR)

SUMMARY:
This study investigates the effects of intensive, high dosage task and impairment based training of the hemiparetic hand, using haptic robots integrated with complex gaming and virtual reality simulations. There is a time-limited period of post-ischemic heightened neuronal plasticity during which intensive training may optimally affect the recovery of motor skills, indicating that the timing of rehabilitation is as important as the dosing. However, recent literature indicates a controversy regarding both the value of intensive, high dosage as well as the optimal timing for therapy in the first two months after stroke. This study is designed to empirically investigate this controversy. It is evident that providing additional, intensive therapy during the acute rehabilitation stay is more complicated to implement and difficult for patients to tolerate, than initiating it in the outpatient setting, immediately after discharge. The robotic/VR system is specifically designed to deliver hand and arm training when motion and strength are limited, using adaptive algorithms to drive individual finger movement, gain adaptation and workspace modification to increase finger and arm range of motion, and haptic and visual feedback from mirrored movements to reinforce motor networks in the lesioned hemisphere.

DETAILED DESCRIPTION:
This study investigates the effects of high dosage task and impairment based training of the hemiparetic hand, using haptic robots integrated with complex gaming and virtual reality simulations on recovery and function of the hand, when the training is initiated within early period of heightened plasticity. The intervention uses two training systems. NJIT-RAVR consists of a data glove combined with the Haptic Master robot that provides tracking of movements in a 3D workspace and enables programmable haptic effects, such as variable anti-gravity support, springs and dampers, and various haptic objects. The NJIT-TrackGlove consists of a robotic hand exoskeleton to provide haptic effects or assistance and an instrumented glove for finger angle tracking, and an arm tracking system to track hand and arm position and orientation. Using programmable software and custom bracing we enable use of this system for patients with a broad set of impairments and functional abilities. A library of custom-designed impairment and task-based simulations that train arm transport and hand manipulation, together or separately will be used. Pilot data show that it is possible to integrate intensive, high-dosage, targeted hand therapy into the routine of an acute rehabilitation setting. The study integrates the behavioral, the kinematic/kinetic and neurophysiological aspects of recovery to determine: 1) whether early intensive training focusing on the hand will result in a more functional hemiparetic arm; (2) whether it is necessary to initiate intensive hand therapy during the very early inpatient rehabilitation phase or will comparable outcomes be achieved if the therapy is initiated right after discharge, in the outpatient period; and 3) whether the effect of the early intervention observed at 6 months post stroke can be predicted by the cortical reorganization evaluated immediately prior to the therapy. This study will fill critical gaps in the literature and make a significant advancement in the investigation of putative interventions for recovery of hand function in patients post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* unilateral right or left sided stroke within 7 to 30 days of starting study
* sufficient cognitive function to follow instructions
* Fugl-Meyer (FM) of ≤ 49/66
* intact cutaneous sensation (e.g. ability to detect <4.17 N stimulation using Semmes- Weinstein nylon filaments

Exclusion Criteria:

* prior stroke with persistent motor impairment or other disabling neurologic condition
* non-independent before stroke
* receptive aphasia
* hemispatial neglect or severe proprioceptive loss
* significant illnesses
* severe arthritis that limits arm and hand movements
* a score of ≥1 on the NIHSS limb ataxia item

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | 4 months post stroke
  The ARAT assesses upper extremity activity. It is a 19 item test divided into four subscales: grasp, grip, pinch and movement. Scores range from 0-57 with higher scores indicating better performance.

SECONDARY OUTCOMES:
Action Research Arm Test | 6 months post stroke
  The ARAT assesses upper extremity activity. It is a 19 item test divided into four
Action Research Arm Test | 1 month post treatment
  The ARAT assesses upper extremity activity. It is a 19 item test divided into four
Action Research Arm Test | Immediately post treatment (ideally within 72 hours)
  The ARAT assesses upper extremity activity. It is a 19 item test divided into four
Action Research Arm Test | Immediately prior to treatment (ideally within 72 hours)
  The ARAT assesses upper extremity activity. It is a 19 item test divided into four
Cortical Area Representation of the Finger-Hand Muscles | 4 months post stroke
  Single-pulse transcranial magnetic stimulation will be used to assay patterns of corticospinal reorganization. Changes in the ipsilesional hand cortical territory for all subjects will be quantified using motor evoked potentials. The topographic representation of the hand and arm muscles will be mapped.
Cortical Area Representation of the Finger-Hand Muscles | 6 months post stroke
  Single-pulse transcranial magnetic stimulation will be used to assay patterns of corticospinal reorganization. Changes in the ipsilesional hand cortical territory for all subjects will be quantified using motor evoked potentials. The topographic representation of the hand and arm muscles will be mapped.
Cortical Area Representation of the Finger-Hand Muscles | 1 month post treatment
  Single-pulse transcranial magnetic stimulation will be used to assay patterns of corticospinal reorganization. Changes in the ipsilesional hand cortical territory for all subjects will be quantified using motor evoked potentials. The topographic representation of the hand and arm muscles will be mapped.
Cortical Area Representation of the Finger-Hand Muscles | Immediately post treatment (ideally within 72 hours)
  Single-pulse transcranial magnetic stimulation will be used to assay patterns of corticospinal reorganization. Changes in the ipsilesional hand cortical territory for all subjects will be quantified using motor evoked potentials. The topographic representation of the hand and arm muscles will be mapped.
Cortical Area Representation of the Finger-Hand Muscles | Immediately prior to treatment (ideally within 72 hours)
  Single-pulse transcranial magnetic stimulation will be used to assay patterns of corticospinal reorganization. Changes in the ipsilesional hand cortical territory for all subjects will be quantified using motor evoked potentials. The topographic representation of the hand and arm muscles will be mapped.
EEG-Based Measure of Resting State Brain Connectivity | 4 months post stroke
  Electroencephalography will be used to evaluate resting-state brain connectivity.
EEG-Based Measure of Resting State Brain Connectivity | 6 months post stroke
  Electroencephalography will be used to evaluate resting-state brain connectivity.
EEG-Based Measure of Resting State Brain Connectivity | 1 month post treatment
  Electroencephalography will be used to evaluate resting-state brain connectivity.
EEG-Based Measure of Resting State Brain Connectivity | Immediately post treatment (ideally within 72 hours)
  Electroencephalography will be used to evaluate resting-state brain connectivity.
EEG-Based Measure of Resting State Brain Connectivity | Immediately prior to treatment (ideally within 72 hours)
  Electroencephalography will be used to evaluate resting-state brain connectivity.
EEG-Based Measure of Task-Based Brain Connectivity | 4 months post stroke
  Task-based connectivity will be evaluated.
EEG-Based Measure of Task-Based Brain Connectivity | 6 months post stroke
  Electroencephalography will be used to evaluate task-based brain connectivity.
EEG-Based Measure of Task-Based Brain Connectivity | 1 month post treatment
  Electroencephalography will be used to evaluate task-based brain connectivity.
EEG-Based Measure of Task-Based Brain Connectivity | Immediately post treatment (ideally within 72 hours)
  Electroencephalography will be used to evaluate task-based brain connectivity.
EEG-Based Measure of Task-Based Brain Connectivity | Immediately prior to treatment (ideally within 72 hours)
  Electroencephalography will be used to evaluate task-based brain connectivity.
Cerebral Oxygenation in Sensorimotor Cortex | 4 months post stroke
  Functional near-infrared spectroscopy will be used to quantify cerebral oxygenation in the sensorimotor cortex during a simple motor task.
Cerebral Oxygenation in Sensorimotor Cortex | 6 months post stroke
  Functional near-infrared spectroscopy will be used to quantify cerebral oxygenation in the sensorimotor cortex during a simple motor task.
Cerebral Oxygenation in Sensorimotor Cortex | 1 month post treatment
  Functional near-infrared spectroscopy will be used to quantify cerebral oxygenation in the sensorimotor cortex during a simple motor task.
Cerebral Oxygenation in Sensorimotor Cortex | Immediately post treatment (ideally within 72 hours)
  Functional near-infrared spectroscopy will be used to quantify cerebral oxygenation in the sensorimotor cortex during a simple motor task.
Cerebral Oxygenation in Sensorimotor Cortex | Immediately prior to treatment (ideally within 72 hours)
  Functional near-infrared spectroscopy will be used to quantify cerebral oxygenation in the sensorimotor cortex during a simple motor task.
Blocks and Box Test | 4 months post stroke
  A unilateral test of manual dexterity scored as the maximum number of blocks that can be moved from one compartment of the box to another of equal size, within 60 seconds.
Blocks and Box Test | 6 months post stroke
  A unilateral test of manual dexterity scored as the maximum number of blocks that can be moved from one compartment of the box to another of equal size, within 60 seconds.
Blocks and Box Test | 1 month post treatment
  A unilateral test of manual dexterity scored as the maximum number of blocks that can be moved from one compartment of the box to another of equal size, within 60 seconds.
Blocks and Box Test | Immediately post treatment (ideally within 72 hours)
  A unilateral test of manual dexterity scored as the maximum number of blocks that can be moved from one compartment of the box to another of equal size, within 60 seconds.
Blocks and Box Test | Immediately prior to treatment (ideally within 72 hours)
  A unilateral test of manual dexterity scored as the maximum number of blocks that can be moved from one compartment of the box to another of equal size, within 60 seconds.
Fugl-Meyer Test of Sensorimotor Function After Stroke (UEFM) | 4 months post stroke
  An impairment based measure consisting of 33 movements that tests motor and sensation of the affected arm. Higher scores indicate less impairment and more isolated motions.
Fugl-Meyer Test of Sensorimotor Function After Stroke (UEFM) | 6 months post stroke
  An impairment based measure consisting of 33 movements that tests motor and sensation of the affected arm. Higher scores indicate less impairment and more isolated motions.
Fugl-Meyer Test of Sensorimotor Function After Stroke (UEFM) | 1 month post treatment
  An impairment based measure consisting of 33 movements that tests motor and sensation of the affected arm. Higher scores indicate less impairment and more isolated motions.
Fugl-Meyer Test of Sensorimotor Function After Stroke (UEFM) | Immediately post treatment (ideally within 72 hours)
  An impairment based measure consisting of 33 movements that tests motor and sensation of the affected arm. Higher scores indicate less impairment and more isolated motions.
Fugl-Meyer Test of Sensorimotor Function After Stroke (UEFM) | Immediately prior to treatment (ideally within 72 hours)
  An impairment based measure consisting of 33 movements that tests motor and sensation of the affected arm. Higher scores indicate less impairment and more isolated motions.
Wolf Motor Function Test | 4 months post stroke
  A 15 item timed test of arm and hand use in patients post stroke. The items begin with simple proximal movements and progress to more complex distal hand movements.
Wolf Motor Function Test | 6 months post stroke
  A 15 item timed test of arm and hand use in patients post stroke. The items begin with simple proximal movements and progress to more complex distal hand movements.
Wolf Motor Function Test | 1 month post treatment
  A 15 item timed test of arm and hand use in patients post stroke. The items begin with simple proximal movements and progress to more complex distal hand movements.
Wolf Motor Function Test | Immediately post treatment (ideally within 72 hours)
  A 15 item timed test of arm and hand use in patients post stroke. The items begin with simple proximal movements and progress to more complex distal hand movements.
Wolf Motor Function Test | Immediately prior to treatment (ideally within 72 hours)
  A 15 item timed test of arm and hand use in patients post stroke. The items begin with simple proximal movements and progress to more complex distal hand movements.
Coordination between Hand Transport and Grasp during Reaching | 4 months post stroke
  The real-world Reach-Grasp test measures the kinematics of everyday movements involving grasping and manipulating household objects. Kinematics of reaching for an object, lifting it from the support, transporting it to a predefined location and releasing the object will be evaluated. Coordination between hand transport and grasping will be evaluated by analyzing hand preshaping during reach.
Coordination between Hand Transport and Grasp during Reaching | 6 months post stroke
  The real-world Reach-Grasp test measures the kinematics of everyday movements involving grasping and manipulating household objects. Kinematics of reaching for an object, lifting it from the support, transporting it to a predefined location and releasing the object will be evaluated. Coordination between hand transport and grasping will be evaluated by analyzing hand preshaping during reach.
Coordination between Hand Transport and Grasp during Reaching | 1 month post treatment
  The real-world Reach-Grasp test measures the kinematics of everyday movements involving grasping and manipulating household objects. Kinematics of reaching for an object, lifting it from the support, transporting it to a predefined location and releasing the object will be evaluated. Coordination between hand transport and grasping will be evaluated by analyzing hand preshaping during reach.
Coordination between Hand Transport and Grasp during Reaching | Immediately post treatment (ideally within 72 hours)
  The real-world Reach-Grasp test measures the kinematics of everyday movements involving grasping and manipulating household objects. Kinematics of reaching for an object, lifting it from the support, transporting it to a predefined location and releasing the object will be evaluated. Coordination between hand transport and grasping will be evaluated by analyzing hand preshaping during reach.
Coordination between Hand Transport and Grasp during Reaching | Immediately prior to treatment (ideally within 72 hours)
  The real-world Reach-Grasp test measures the kinematics of everyday movements involving grasping and manipulating household objects. Kinematics of reaching for an object, lifting it from the support, transporting it to a predefined location and releasing the object will be evaluated. Coordination between hand transport and grasping will be evaluated by analyzing hand preshaping during reach.
Arm Range of Motion | 4 months post stroke
  Active range of motion for fingers, wrist, elbow and shoulder.
Arm Range of Motion | 6 months post stroke
  Active range of motion for fingers, wrist, elbow and shoulder.
Arm Range of Motion | 1 month post treatment
  Active range of motion for fingers, wrist, elbow and shoulder.
Arm Range of Motion | Immediately post treatment (ideally within 72 hours)
  Active range of motion for fingers, wrist, elbow and shoulder.
Arm Range of Motion | Immediately prior to treatment (ideally within 72 hours)
  Active range of motion for fingers, wrist, elbow and shoulder.
Accuracy of Tracking a Square and Sine Wave with Fingertip Pinch Force | 4 months post stroke
  Ability to regulate force will be evaluated by measuring the accuracy of tracking square and sine waves presented on a computer screen. Vertical position of the cursor on the screen will be defined by isometric force between the thumb and index fingertips measured by a force sensor.
Accuracy of Tracking a Square and Sine Wave with Fingertip Pinch Force | 6 months post stroke
  Ability to regulate force will be evaluated by measuring the accuracy of tracking square and sine waves presented on a computer screen. Vertical position of the cursor on the screen will be defined by isometric force between the thumb and index fingertips measured by a force sensor.
Accuracy of Tracking a Square and Sine Wave with Fingertip Pinch Force | 1 month post treatment
  Ability to regulate force will be evaluated by measuring the accuracy of tracking square and sine waves presented on a computer screen. Vertical position of the cursor on the screen will be defined by isometric force between the thumb and index fingertips measured by a force sensor.
Accuracy of Tracking a Square and Sine Wave with Fingertip Pinch Force | Immediately post treatment (ideally within 72 hours)
  Ability to regulate force will be evaluated by measuring the accuracy of tracking square and sine waves presented on a computer screen. Vertical position of the cursor on the screen will be defined by isometric force between the thumb and index fingertips measured by a force sensor.
Accuracy of Tracking a Square and Sine Wave with Fingertip Pinch Force | Immediately prior to treatment (ideally within 72 hours)
  Ability to regulate force will be evaluated by measuring the accuracy of tracking square and sine waves presented on a computer screen. Vertical position of the cursor on the screen will be defined by isometric force between the thumb and index fingertips measured by a force sensor.
Maximum Thumb and Index Fingertip Pinch Force | 4 months post stroke
  A force sensor will be used to measure in Newtons maximum isometric pinch force achieved between the thumb and index fingertips.
Maximum Thumb and Index Fingertip Pinch Force | 6 months post stroke
  A force sensor will be used to measure in Newtons maximum isometric pinch force achieved between the thumb and index fingertips.
Maximum Thumb and Index Fingertip Pinch Force | 1 month post treatment
  A force sensor will be used to measure in Newtons maximum isometric pinch force achieved between the thumb and index fingertips.
Maximum Thumb and Index Fingertip Pinch Force | Immediately post treatment (ideally within 72 hours)
  A force sensor will be used to measure in Newtons maximum isometric pinch force achieved between the thumb and index fingertips.
Maximum Thumb and Index Fingertip Pinch Force | Immediately prior to treatment (ideally within 72 hours)
  A force sensor will be used to measure in Newtons maximum isometric pinch force achieved between the thumb and index fingertips.
Accuracy of Tracking a Square and Sine Wave with Isotonic Finger Flexion/Extension | 4 months post stroke
  A data glove will be used to evaluate the accuracy of tracking square and sine waves presented on a computer screen with isotonic finger flexion/extension. Vertical position of the cursor on the screen will be defined by the average of four metacarpophalangeal finger joints.
Accuracy of Tracking a Square and Sine Wave with Isotonic Finger Flexion/Extension | 6 months post stroke
  A data glove will be used to evaluate the accuracy of tracking square and sine waves presented on a computer screen with isotonic finger flexion/extension. Vertical position of the cursor on the screen will be defined by the average of four metacarpophalangeal finger joints.
Accuracy of Tracking a Square and Sine Wave with Isotonic Finger Flexion/Extension | 1 month post treatment
  A data glove will be used to evaluate the accuracy of tracking square and sine waves presented on a computer screen with isotonic finger flexion/extension. Vertical position of the cursor on the screen will be defined by the average of four metacarpophalangeal finger joints.
Accuracy of Tracking a Square and Sine Wave with Isotonic Finger Flexion/Extension | Immediately post treatment (ideally within 72 hours)
  A data glove will be used to evaluate the accuracy of tracking square and sine waves presented on a computer screen with isotonic finger flexion/extension. Vertical position of the cursor on the screen will be defined by the average of four metacarpophalangeal finger joints.
Accuracy of Tracking a Square and Sine Wave with Isotonic Finger Flexion/Extension | Immediately prior to treatment (ideally within 72 hours)
  A data glove will be used to evaluate the accuracy of tracking square and sine waves presented on a computer screen with isotonic finger flexion/extension. Vertical position of the cursor on the screen will be defined by the average of four metacarpophalangeal finger joints.
Measurement of Daily Use of Upper Extremity | 4 months post stroke
  Wearable sensors will be used to quantify daily use of the affected arm after the intervention.
Measurement of Daily Use of Upper Extremity | 6 months post stroke
  Wearable sensors will be used to quantify daily use of the affected arm after the intervention.
Measurement of Daily Use of Upper Extremity | 1 month post treatment
  Wearable sensors will be used to quantify daily use of the affected arm after the intervention.
EuroQol | 4 months post stroke
  The EuroQol - EQ-5D is a standardized instrument used as a measure of health-related quality of life. The descriptive system comprises five dimensions: 1. mobility, the person's walking ability; 2. self-care, the ability to wash or dress by oneself; 3. usual activities dimension, performance in "work, study, housework, family or leisure activities"; 4. pain/discomfort, how much pain or discomfort they have, and 5. anxiety/depression, how much anxious or depressed they are. The respondents self-rate their level of severity for each dimension.
EuroQol | 6 months post stroke
  The EuroQol - EQ-5D is a standardized instrument used as a measure of health-related quality of life. The descriptive system comprises five dimensions: 1. mobility, the person's walking ability; 2. self-care, the ability to wash or dress by oneself; 3. usual activities dimension, performance in "work, study, housework, family or leisure activities"; 4. pain/discomfort, how much pain or discomfort they have, and 5. anxiety/depression, how much anxious or depressed they are. The respondents self-rate their level of severity for each dimension.
EuroQol | 1 month post treatment
  The EuroQol - EQ-5D is a standardized instrument used as a measure of health-related quality of life. The descriptive system comprises five dimensions: 1. mobility, the person's walking ability; 2. self-care, the ability to wash or dress by oneself; 3. usual activities dimension, performance in "work, study, housework, family or leisure activities"; 4. pain/discomfort, how much pain or discomfort they have, and 5. anxiety/depression, how much anxious or depressed they are. The respondents self-rate their level of severity for each dimension.
EuroQol | Immediately post treatment (ideally within 72 hours)
  The EuroQol - EQ-5D is a standardized instrument used as a measure of health-related quality of life. The descriptive system comprises five dimensions: 1. mobility, the person's walking ability; 2. self-care, the ability to wash or dress by oneself; 3. usual activities dimension, performance in "work, study, housework, family or leisure activities"; 4. pain/discomfort, how much pain or discomfort they have, and 5. anxiety/depression, how much anxious or depressed they are. The respondents self-rate their level of severity for each dimension.
EuroQol | Immediately prior to treatment (ideally within 72 hours)
  The EuroQol - EQ-5D is a standardized instrument used as a measure of health-related quality of life. The descriptive system comprises five dimensions: 1. mobility, the person's walking ability; 2. self-care, the ability to wash or dress by oneself; 3. usual activities dimension, performance in "work, study, housework, family or leisure activities"; 4. pain/discomfort, how much pain or discomfort they have, and 5. anxiety/depression, how much anxious or depressed they are. The respondents self-rate their level of severity for each dimension.
National Institutes of Health Stroke Scale (NIHSS) | 4 months post stroke
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate and document neurological status in stroke patients and the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3 to 5 grades with 0 as normal.
National Institutes of Health Stroke Scale (NIHSS) | 6 months post stroke
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate and document neurological status in stroke patients and the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3 to 5 grades with 0 as normal.
National Institutes of Health Stroke Scale (NIHSS) | 1 month post treatment
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate and document neurological status in stroke patients and the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3 to 5 grades with 0 as normal.
National Institutes of Health Stroke Scale (NIHSS) | Immediately post treatment (ideally within 72 hours)
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate and document neurological status in stroke patients and the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3 to 5 grades with 0 as normal.
National Institutes of Health Stroke Scale (NIHSS) | Immediately prior to treatment (ideally within 72 hours)
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate and document neurological status in stroke patients and the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3 to 5 grades with 0 as normal.
Change in Robot-Based Measure of Elbow-Shoulder Coordination during Reaching | Day 1 and and Day 10 of treatment for EVR and DVR groups
  To compare the immediate effects of training in the EVR and DVR groups, subjects will reach to five haptically rendered spheres located in a 3D virtual environment. The test will be performed every day immediately prior to VR training to measure changes in patterns of elbow-shoulder coordination.
Change in Robot-Based Measure of Maximum Seated Workspace during Reaching | Day 1 and and Day 10 of treatment for EVR and DVR groups
  To compare the immediate effects of training in the EVR and DVR groups, subjects will reach to five haptically rendered spheres located in a 3D virtual environment. The test will be performed every day immediately prior to VR training to measure changes in maximum seated workspace.
Change in Robot-Based Measure of Movement Speed during Arm Reaching | Day 1 and and Day 10 of treatment for EVR and DVR groups
  To compare the immediate effects of training in the EVR and DVR groups, subjects will reach to five haptically rendered spheres located in a 3D virtual environment. The test will be performed immediately prior to VR training to measure changes in arm speed during reaching for a virtual target.
Change in Robot-Based Measure of Movement Speed during Targeted Finger Motion | Day 1 and and Day 10 of treatment for EVR and DVR groups
  To compare the immediate effects of training in the EVR and DVR groups, subjects will perform targeted finger movements in a virtual environment. The test will be performed every day immediately prior to VR training to measure changes in the speed of finger movement towards a virtual target.
Patient's Structured Subjective Assessment | Immediately post treatment (ideally within 72 hours) for EVR and DVR groups
  This is a 27 item questionnaire that addresses the subjects perception of the function of their hemiplegic arm and the effect this intervention had on their hand function. Subjects fill out the questionnaire prior to and directly after the intervention. Some questions require a response such as disagree, neutral and agree, others require ordering their gaming activity preferences, or responding to a question with a short answer.

CONTACTS AND LOCATIONS:
Overall Officials: Sergei V Adamovich, PhD, Principal Investigator — New Jersey Institute of Technology; Alma S Merians, PhD, PT, Principal Investigator — Rutgers University; Karen Nolan, PhD, Principal Investigator — Kessler Foundation; Eugene Tunik, PhD, PT, Principal Investigator — Northeastern University
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, Saddle Brook, New Jersey
  - Kessler Institute for Rehabilitation, West Orange, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Merians AS, Fluet GG, Qiu Q, Yarossi M, Patel J, Mont AJ, Saleh S, Nolan KJ, Barrett AM, Tunik E, Adamovich SV. Hand Focused Upper Extremity Rehabilitation in the Subacute Phase Post-stroke Using Interactive Virtual Environments. Front Neurol. 2020 Nov 26;11:573642. doi: 10.3389/fneur.2020.573642. eCollection 2020. PMID 33324323